CLINICAL TRIAL: NCT06015282
Title: A Phase 3, Randomized, Observer-Blind, Controlled, Multicenter, Clinical Study to Evaluate Immunogenicity and Safety of a MF59-Adjuvanted Quadrivalent Subunit Cell-derived Influenza Vaccine (aQIVc) in Comparison With Quadrivalent Influenza Vaccines, in Adults Aged 50 Years and Older.
Brief Title: The Celljuvant Study: A Phase 3 Immunogenicity and Safety Study of aQIVc Vaccine in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V201_03
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Influenza, Human
Keywords: influenza; vaccine; MF59; Adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational aQIVc group (Experimental)
  Interventions: Biological: Investigational aQIVc
- licensed QIVr group (Active Comparator)
  Interventions: Biological: licensed QIVr
- licensed aQIV group (Active Comparator)
  Interventions: Biological: licensed aQIV

INTERVENTIONS:
Biological: Investigational aQIVc — Investigational Adjuvanted Cell-derived Quadrivalent Influenza vaccine, containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO (World Health Organization) for quadrivalent vaccines for the respective season.
  Arms: Investigational aQIVc group
Biological: licensed QIVr — Recombinant Quadrivalent Influenza Vaccine (Flublok Quadrivalent/Supemtek) containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO for quadrivalent vaccines for the respective season.
  Arms: licensed QIVr group
Biological: licensed aQIV — Adjuvanted, egg-derived Quadrivalent Influenza Vaccine (Fluad) containing four influenza virus strains (A/H1N1, A/H3N2, B/Yamagata and Victoria lineage) recommended by the WHO for quadrivalent vaccines for the respective season.
  Arms: licensed aQIV group

SUMMARY:
This is a Phase 3, randomized, parallel-group, comparator-controlled, observer-blind, multicenter study of immunogenicity and safety in approximately 7700 male and female adults aged 50 years and older (approximately equally split between two age groups: 50-64 years; 65 years and older), who are healthy or have stable comorbidities that increase their risk of complications from influenza infection. Three lots of aQIVc will be evaluated for consistency and pooled for the comparison with the 2 control vaccines.

Subjects will be randomly assigned to receive 1 of 3 lots of aQIVc, QIVr, or aQIV in a 1:1:1:2:2 ratio (for a 3:2:2 ratio for aQIVc, QIVr, and aQIV).

The study will have a treatment period (Day 1 to Day 29) and a follow-up period (Day 30 up to Day 181); a subset of 770 subjects will be followed up up to Day 365.

ELIGIBILITY:
Main Inclusion Criteria:

* Individuals, aged 50 years and older, who are healthy or have stable comorbidities that increase their risk of complications from influenza infection
* Individuals who can comply with all study procedures

Main Exclusion Criteria:

* Progressive, unstable, or uncontrolled clinical conditions
* Known hypersensitivity or allergy to any study vaccine component
* Known history of Guillain-Barré syndrome or other demyelinating disease
* Condition representing a contraindication to vaccination or blood draw
* Abnormal function of immune system due to known disorder or medication.
* Influenza vaccination within 180 days prior to informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7741 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Immunogenicity Endpoint: Humoral immune responses of 3 lots of aQIVc compared in pairs in terms of Day 29 GMT ratio between each pair among the 3 lots, from antibody titers measured via HI assay. | Day 29
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains.
Immunogenicity Endpoint: Humoral immune responses of aQIVc in comparison with QIVr and aQIV vaccines in terms of Day 29 GMT and GMT ratio of antibodies measured via HI assay. | Day 29
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains.
  Noninferiority of aQIVc versus comparator (QIVr or aQIV) will be demonstrated if the lower limit (LL) of the 2-sided 97.5% CI for the Day 29 GMT ratio (aQIVc/comparator) is ≥0.67 for each of the 4 vaccine strains.
Immunogenicity Endpoint: Humoral immune responses of aQIVc in comparison with QIVr and aQIV vaccines in terms of Day 1 to Day 29 SCR and SCR difference, from antibody titers measured via HI assay. | Day 1 and Day 29
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains.
  SCR is the percentage of subjects with seroconversion (defined as either a prevaccination [Day 1] titer <1:10 and a postvaccination [Day 29] titer ≥1:40, or a prevaccination titer ≥1:10 and a ≥4-fold increase in postvaccination titer).
  Noninferiority of aQIVc versus comparator (QIVr or aQIV) will be demonstrated if the lower limit (LL) of the 2-sided 97.5% CI for the difference in SCR (aQIVc minus comparator) is ≥-10% for each of the 4 vaccine strains.

SECONDARY OUTCOMES:
Immunogenicity Endpoint: Humoral immune responses of aQIVc in comparison with aQIV vaccine in terms of Day 29 SCR and SCR difference, GMT and GMT ratio of antibodies measured via HI assay in subjects 65 years and older. | Day 1 and Day 29
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains.
  Noninferiority will be demonstrated if the LL of the 2-sided adjusted CI for the Day 29 GMT ratio (aQIVc/comparator) is ≥0.67 for each of the 4 vaccine strains, and the LL of the 2-sided adjusted CI for the difference in SCR (aQIVc minus comparator) is ≥-10% for each of the 4 vaccine strains.
Immunogenicity Endpoint: Humoral immune responses of aQIVc in comparison with QIVr and aQIV vaccines in terms of Day 29 GMT and GMT ratio of antibodies measured via HI assay. | Day 29
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains.
  Superiority of aQIVc versus comparator (QIVr and aQIV) will be demonstrated if the LL of the 2-sided 97.5% CI for the inter-group GMT ratio (aQIVc/comparator) is >1.0 for each of the 4 vaccine strains.
Immunogenicity Endpoints: For aQIVc, QIVr, and aQIV vaccines, Day 29 GMT, Day 1 to Day 29 GMFI, Percentage of subjects with HI titer ≥1:40 at Day 29, Day 1 to Day 29 SCR, SCR differences and GMT ratio of antibodies measured via HI assay. | Day 1 and Day 29
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains, overall and by age subgroup.
Immunogenicity Endpoints: For aQIVc and aQIV vaccines, Day 29 GMT, Day 1 to Day 29 GMFI, Percentage of subjects with HI titer ≥1:40 at Day 29, Day 1 to Day 29 SCR, SCR differences, and GMT ratio of antibodies measured via HI assay. | Day 1 and Day 29
  HI assay will be measured using egg-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains in the HI-egg subset of 2750 subjects, overall and by age subgroup.
Immunogenicity Endpoints: For aQIVc, QIVr and aQIV vaccines, GMT, GMFI, Percentage of subjects with HI titer ≥1:40, SCR, SCR differences, and GMT ratio of antibodies measured via HI assay. | Day 1 up to Day 365
  HI assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains in the long-term subset of 770 subjects, overall and by age subgroup.
Immunogenicity Endpoints: For aQIVc, QIVr and aQIV vaccines, GMT, GMFI, SCR, SCR difference, and GMT ratio of antibodies measured via MN assay. | Day 1 up to Day 365
  MN assay will be measured using cell-derived target viruses for the A/H1N1, A/H3N2, B/Yamagata, and B/Victoria vaccine strains in the long-term subset of 770 subjects, overall and by age subgroup.
Safety endpoints: For aQIVc, QIVr and aQIV vaccines, the percentages of Subjects with Solicited Local Adverse Events, Solicited Systemic Adverse Events, and Severe Solicited Local and/or Systemic AEs. | Day 1 to Day 7
Safety endpoints: For aQIVc, QIVr and aQIV vaccines, the percentage of Subjects with Unsolicited Adverse Events. | Day 1 to Day 29
Safety endpoints: For aQIVc, QIVr and aQIV vaccines, the percentages of subjects with Serious Adverse Events (SAEs), AEs Leading to Withdrawal, Adverse Events of Special Interest (AESI) and non-serious Medically Attended Adverse Events (MAAEs). | Day 1 to Day 181
Safety endpoints: For aQIVc, QIVr and aQIV vaccines, the percentages of subjects with Serious Adverse Events (SAEs), AEs Leading to Withdrawal, Adverse Events of Special Interest (AESI) and non-serious Medically Attended Adverse Events (MAAEs). | Day 1 to Day 365
  Long-term safety for the long-term subset of 770 subjects

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (96):
- United States (51):
  - Alliance for Multispecialty Research (AMR) Phoenix, Tempe, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Marvel Clinical Research, Huntington Beach, California
  - Paradigm Clinical Research Center, LLC, Redding, California
  - Clinical Research Consulting, Inc., Milford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - USA and International Research Inc., Doral, Florida
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - ARS - Lake Oconee, Largo, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Global Health Research center, Tampa, Florida
  - Velocity Clinical Research- Boise, Meridian, Idaho
  - Great Lakes Clinical Trials, LLC Ravenswood dba Flourish Research, Chicago, Illinois
  - Great Lakes Clinical Trials, LLC. Ravenswood dba Flourish Research, Gurnee, Illinois
  - Velocity Clinical Research Valparaoso, Valparaiso, Indiana
  - Velocity Clinical Research, Sioux City, Sioux City, Iowa
  - Velocity Clinical Research, Baton Rough, Baton Rouge, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - IMA Evaluations LLC, Monroe, Louisiana
  - Centennial Medical Group, PC, Columbia, Maryland
  - Velocity Clinical Research Rockville, Rockville, Maryland
  - Velocity Clinical Research Gulfport, Gulfport, Mississippi
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Alliance for Multispecialty Research (AMR) LLC, Las Vegas, Las Vegas, Nevada
  - Velocity Clinical Research, Binghamton, Binghamton, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - Velocity Clinical Research, Vestal, New York, New York
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Velocity Clinical Research, Spartanburg, Spartanburg, South Carolina
  - AMR-Knoxville, Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Cedar Health Research, LLC, Dallas, Texas
  - Benchmark Research, Fort Worth, Texas
  - DM Clinical Research - Martin Diagnostic Clinic, Houston, Texas
  - ACRC trials Parent HQ, Plano, Texas
  - DM Clinical Research, Tomball, Texas
  - BBCR Holdings LLC dba JBR Clinical Research - Midvale Campus, Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Velocity Clinical Research, Suffolk, Suffolk, Virginia
- CARe Clinic, Red Deer, Alberta, Canada
- Denmark (2):
  - Amager-Hvidovre Hospital, Hvidovre
  - Zealand University Hospital, Roskilde, Roskilde
- Estonia (7):
  - Vee Family Doctor's Center OY, Paide
  - OÜ Innomedica, Tallinn
  - Center for Clinical and Basic Research, Tallinn
  - Al Mare Perearstikeskus OÜ, Tallinn
  - Merelahe Family Doctors Centre, Tallinn
  - Clinical Research Centre, Tartu
  - Tartu University Hospital, Tartu
- Germany (16):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - emovis GmbH, Berlin
  - Velocity Clinical Research, Berlin, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Klinisches Forschungszentrum Dr. Hagemann am Hausarztzentrum am Germaniaplatz Dr.Hagemann/ Breider, Essen
  - Studienzentrum Bocholderstrasse, Essen
  - UHZ Klinische Forschung, Essen
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Velocity Clinical Research, Hamburg, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Velocity Clinical Research, Leipzig, Leipzig
  - Studienzentrum FMZ Radowsky, Leipzig
  - Research Quist, Mainz
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Studienzentrum Leitz Triderm, Stuttgart
- Pakistan (2):
  - The Aga Khan University, Karachi
  - Central Park Teaching Hospital, Lahore
- Philippines (12):
  - Silang Specialists Medical Center, Silang, Cavite
  - Davao Medical School Foundation Inc. Hospital / NEMESIO F. ANLOCOTAN III, Davao City, Davao Del Sur
  - Las Pinas Doctors Hospital, Las Piñas, Las Pinas City
  - Marilao Saint Michael Family Hospital, Inc, Bulacan
  - CARE CT Group Inc. CARE Clinical Trials, Cavite
  - Health Index Multispecialty and Lying in Clinic, Cavite
  - Norzel Medical and Diagnostic Clinic, Cebu City
  - Ospital ng Makati, City of Taguig
  - West Visayas State University Medical Center, Iloilo City
  - Manila Doctors Hospital, Manila
  - Mary Johnston Hospital, Manila
  - Quirino Memorial Medical Center, Quezon City
- United Kingdom (5):
  - Velocity High Wycombe, High Wycombe
  - Velocity North London, London
  - Panthera Biopartners Ltd (Preston), Preston
  - Panthera Biopartners Ltd (Manchester), Rochdale
  - Panthera Biopartners (Sheffield), Sheffield

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the Common Technical Document (CTD) modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])).
Supporting Information: Study Protocol, SAP
Time Frame: SEQIRUS discloses results from clinical studies within 12 months of last patient last visit (LPLV) unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication.
URL: https://www.seqirus.us/partnering